CLINICAL TRIAL: NCT01121458
Title: Clevidipine for Vasoreactivity Evaluation of the Pulmonary Arterial Bed (CARVE)
Brief Title: Clevidipine for Vasoreactivity Evaluation of the Pulmonary Arterial Bed
Acronym: CARVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Chief- Division of Cardiology, North Texas Veterans Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dallas VA #09-041
Record Dates: First submitted 2010-02-02; First posted 2010-05-12 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary artery; vascular resistance
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevidipine — The clevidipine infusion is to be administered via IV infusion at a starting dose of 0.5 mg/hour. The dose may be doubled every three (3) minutes to a maximum dose of 32 mg/hr as tolerated, until a 20% reduction in PVR is achieved or until the patient experiences hypotension (SBP< 80 mmHg), hypertension (SBP>150 mmHg), tachycardia (120 beats per minute), bradycardia (<50 beats per minute), or symptoms of hypotension or ischemia (chest pain, anxiety, nausea, vomiting), allergic reaction (hives, urticaria) or other adverse event. Clevidipine infusion may be terminated at any time for a safety reason or at the investigator's discretion.
  Other Names: Cleviprex

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare blood vessel disorder of the lung in which the pressure in the pulmonary artery (PA) rises above normal levels and may become life threatening. PAH is frequently misdiagnosed and has often progressed to late stage by the time it is accurately diagnosed. PAH has been historically chronic and incurable with a poor survival rate. However, new treatments are available which have significantly improved prognosis. Right-heart catheterization (RHC) is the most accurate and useful test for PAH, and the only test that directly measures the pressure inside the PA. It is performed in all patients at least once, to get a definitive diagnosis of PAH.

The most commonly used medication for this purpose is intravenous nitroprusside, however this medication in about 25-30% of patients is not well tolerated as it cause fast heart rates, which is not well tolerated by patients with pulmonary hypertension and/or heart failure. The CARVE study assesses the effect of Clevidipine, an ultra-short acting vasoselective calcium antagonist, on pulmonary vascular resistance (PVR) and its utility for pulmonary vasoreactivity testing during right heart catheterization (RHC) of patients with pulmonary hypertension (PAH).

DETAILED DESCRIPTION:
CARVE is a Phase 4 open-label descriptive observational trial in PAH patients undergoing invasive vasoreactivity testing in the cath lab at the Dallas VA Medical Center. Patients clinically indicated for RHC and assessment of pulmonary artery vasoreactivity will be enrolled if they meet the inclusion/exclusion criteria. The study will involve the following tests:

1. Performance of clinically indicated RHC with assessment of pulmonary hypertension and pulmonary vascular resistance (PVR).
2. Performance of clinically indicated pulmonary vasoreactivity assessment with IV Nitroprusside (standard of care)
3. For patients who are responsive to Nitroprusside, or those who have an inconclusive result because of intolerability to Nitroprusside, pulmonary vasoreactivity assessment with study drug (IV) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before initiation of any study related procedures.
* 21 years of age or older
* Referred for clinically indicated pulmonary vascular resistance assessment
* Presence of pulmonary hypertension by non-invasive testing
* Patients referred for RHC and vasoreactivity testing

Exclusion Criteria:

* Patient with baseline SBP < 100 mmHg
* Patient with HR>120 beats/minute
* Patients with severe or valvular heart disease
* Patients with an acute coronary syndrome
* Patients with a creatinine clearance < 30 ml/min
* Patients with class IV congestive heart failure
* Patients with platelet count < 100,000 per cc3
* Patients with hemoglobin < 10g/dl
* Patient with INR > 1.5
* Patients with positive pregnancy test - women between 21 and 60 years of age
* Patients with known or suspected allergy to study drug or study drug components, including allergy to soybeans, soy products, eggs, or egg products
* Patients with defective lipid metabolism such as pathologic hyperlipemia, lipoid nephrosis, or acute pancreatitis if it is accompanied by hyperlipidemia
* Patients with contraindications to the use of IV nitroprusside
* Patients with diagnosed or suspected intra-cardiac or systemic arteriovenous shunts
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 3 months of randomization.
* Other medical conditions that, in the opinion of the investigator, preclude participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Percent reduction in PVR with clevidipine in (1) nitroprusside responders and (2) patients with indeterminate nitroprusside reactivity tests | During right heart catheterization (1-2 hours)

SECONDARY OUTCOMES:
Efficacy/ safety measured by % reduction in PVR with clevidipine in patients with indeterminate reactivity tests & total study population;%patients with successful 20% reduction in PVR; SAE & adverse hemodynamic response to clevidipine during procedure | During right heart catheterization (1-2 hrs)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States